CLINICAL TRIAL: NCT06240156
Title: Effect of Insole Intervention on Plantar Pressure Distribution, Gait Balance and Lower Back Pain in Flatfoot Women During the Third Trimester
Brief Title: A Study on Plantar Pressure Distribution, Gait Balance and Lower Back Pain in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wan-Lin Pan, assistant professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-S-023-1
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: pregnancy, gait balance, foot pain, lower back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D arch pad design Insole group (Experimental): This study utilizes a custom-made arch support pad with a 3D three-dimensional design that is already available on the market (patent number I315187). Its arch support principle is designed using 3DBS (Three-Dimensional Biomechanics System - 3DBS), which can conform to the user's feet. In this type, the bottom layer provides an overall shock-absorbing function.
  Interventions: Other: 3D arch pad design Insole group
- flat Insole group (Placebo Comparator): General Insole without any special features
  Interventions: Other: flat Insole group

INTERVENTIONS:
Other: 3D arch pad design Insole group — 3D three-dimensional design that is already available on the market (patent number I315187). Its arch support principle is designed using 3DBS (Three-Dimensional Biomechanics System - 3DBS), which can conform to the user's feet.
  Arms: 3D arch pad design Insole group
Other: flat Insole group — General Insole without any special features
  Arms: flat Insole group

SUMMARY:
The purpose of this study was to understand women with low arched feet, flat feet, or BMI> 29 in the third trimester.

DETAILED DESCRIPTION:
The purpose of this study was to understand women with low arched feet, flat feet, or BMI> 29 in the third trimester. Compare the intervention measures of different foot pads immediately, two weeks, four weeks, and six weeks after the intervention Immediate and long-term benefits in relief of plantar pressure, dynamic and static balance, and lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* able to understand and write Chinese
* health and third trimester women
* low arched feet or flat feet or BMI> 29

Exclusion Criteria:

* Women with a medical record of back, foot, ankle, knee, musculoskeletal, or neuromuscular trauma or disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
plantar pressure | footpad intervention measures immediately, two weeks, four weeks, six weeks after intervention
  The pedar® system, an accurate and reliable pressure distribution measuring system designed to monitor local loads between the foot and the shoe.
static balance | footpad intervention measures immediately, two weeks, four weeks, six weeks after intervention
  The Timed Up and Go (TUG) test is utilized to assess mobility. It is a simple evaluation that measures the speed at which you can stand up, walk 10 feet, turn around, walk back, and sit down.
foot pain | footpad intervention measures immediately, two weeks, four weeks, six weeks after intervention
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning.
lower back pain | footpad intervention measures immediately, two weeks, four weeks, six weeks after intervention
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning.
daily life disturbance scales | footpad intervention measures immediately, two weeks, four weeks, six weeks after intervention
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Meei-Ling Gau, PHD, Principal Investigator — professor
Locations (1):
- Wan-Lin Pan, Taipei, Taiwan